CLINICAL TRIAL: NCT00676377
Title: A New Approach of Neostigmine in Unavoidable Post Operative Ileus After Surgery
Brief Title: A New Approach of Neostigmine in Unavoidable Post Operative Ileus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: S.Ahmad Fanaei,Assistant professor of Surgery, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 8771148z
Record Dates: First submitted 2008-05-12; First posted 2008-05-13 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Ileus
Keywords: Neostigmine, Post Operative, Ileus
MeSH Terms: conditions — Ileus | interventions — Neostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Neostigmine
  Interventions: Drug: Neostigmine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Neostigmine — 2.5 mg of neostigmine intravenously in 250 ml normal saline over a period of thirty minutes ,Half Life 3 Hours
  Other Names: Neostigmine Group
  Arms: 1
Drug: Saline — Saline Placebo
  Other Names: Placebo Group
  Arms: 2

SUMMARY:
Postoperative ileus (POI) in the absence of any mechanical obstruction remains a commonly encountered clinical problem.So, this study aimed to show the effective way to decrease the rate of postoperative Ileus (POI).

DETAILED DESCRIPTION:
We honestly declare that, the use of parasympathomimetic agents such as neostigmine is not without risk. Patients with underlying bradyarrhythmias or those receiving β-adrenergic antagonists may be more susceptible to neostigmine-induced bradycardia. Similarly, neostigmine increases airway secretions and bronchial reactivity, which may exacerbate active bronchospasm. Recently, a new class of drugs-peripherally acting mu-opioid receptor antagonists-may help enhance multimodal management of POI. Although, the cost benefit of the new class of drugs is debated. It has been suggested that the individual components of multimodal protocols-for example, laparoscopy-may reduce certain post surgical morbidities (including POI) But do not by them prevent POI. Therefore, combinations of strategies with demonstrated effectiveness-early feeding , epidural analgesia, laparoscopic surgery, and use of peripherally acting mu-opioid-receptor antagonists-may help transform the reactive approach to POI into a proactive multimodal paradigm that effectively targets the diverse etiologic factors leading to this common clinical problem.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute colonic pseudo-obstruction who were 18 years of age or older
* Patients had to have a cecal diameter of at least 10 cm on plain radiographs
* Mechanical obstruction was ruled out by the finding of air throughout all colonic segments including the rectosigmoid on plain abdominal radiographs

Exclusion Criteria:

* Exclusion criteria included a base-line heart rate of less than 60 beats per minute or systolic blood pressure of less than 90 mm Hg; signs of bowel perforation
* With peritoneal signs on physical examination or free air on radiographs; active bronchospasm requiring medication
* Treatment with prokinetic drugs such as cisapride or metoclopramide in the 24 hours before evaluation
* A history of colon cancer or partial colonic resection
* Active gastrointestinal bleeding
* Pregnancy
* Positive history of Myocardial Infarction, Intestinal Resection or a serum creatinine concentration of more than 3 mg per deciliter (265 µmol per liter)

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
show the effective way to decrease the rate of postoperative Ileus (POI). | 6 hours

SECONDARY OUTCOMES:
abdominal circumference, colonic diameters, and clinical response were again measured. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: S.Ahmad Fanaei, M.D., Study Chair — Baqyiattalah University of Medical Science; S.Ali Ziaee, M.D., Principal Investigator — Erfan Hospital
Locations (1):
- Baqyiattalah University of Medical Science, Tehran, Iran

REFERENCES:
- [Result] Ponec RJ, Saunders MD, Kimmey MB. Neostigmine for the treatment of acute colonic pseudo-obstruction. N Engl J Med. 1999 Jul 15;341(3):137-41. doi: 10.1056/NEJM199907153410301. PMID 10403850